CLINICAL TRIAL: NCT05866939
Title: Development of a Multidisciplinary Network for Clinical and Laboratory Research for Spinal Muscular Atrophy and Other Rare Motoneuron Diseases
Brief Title: Development of a Multidisciplinary Network for Clinical and Laboratory Research for SMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ospedale Pediatrico Bambin Gesù (Other); IRCCS Eugenio Medea (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Other Study IDs: 5496
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to to establish profiles of clinical progression in patients affected by the different types of SMA (type I, II and III) treated with the currently approved drugs using a structured battery of clinical tests.

Another goal of the study is to assess the progression of the disease in patients identified through neonatal screening.

DETAILED DESCRIPTION:
The collection of 2-year longitudinal clinical data will be conducted in newly treated patients at baseline, 6-, 12-, 14- and 22-months post-treatment. Parameters will include motor function, fatigability, respiratory function, event-free survival and death, and swallowing and feeding modalities. It is anticipated that at least 30 new patients will be enrolled in the study.

Importantly, information will also be collected on patients who may decide to switch treatment during the duration of our study, trying to establish if the switch to a new drug (or as an add-on should patients take a new treatment after being treated with gene therapy) may be associated with changes in clinical phenotype.

The aim is to apply a newly established clinical protocol that allows identifying minor signs of disease that are easily missed in the absence of an NBS-detected diagnosis. Indeed, not all infants identified as SMA-positive through the NBS are truly asymptomatic, as a proportion of them may appear paucisymptomatic and their minor signs could be possibly not detected in the absence of a positive screening test.

ELIGIBILITY:
Inclusion Criteria:

* All SMA patients

Exclusion Criteria:

* Inability to understand or to provide informed consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spinal muscular atrophy regardless of age, type of SMA or treatment
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Establish profiles of clinical progression in patients affected by the different types of SMA (type I, II and III) treated with the currently approved drugs using a structured battery of clinical tests. | 2-year
Assess the progression of the disease in patients identified through neonatal screening | 2-year
Identification of molecular biomarkers that associate with disease course and response to therapies | 2-year